CLINICAL TRIAL: NCT06782724
Title: The Safety and Efficacy of Psilocybin Therapy Compared to Low-dose Control in Reducing Depressive Symptoms in Patients with COPD, ALS, MS, or APD.
Brief Title: Psilocybin Therapy for Psychological Distress in Palliative Patients
Acronym: PsyPal
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: HumanKindLabs (Unknown); University of Copenhagen (Other); CTC Clinical Trial Consultants AB (Industry); OPEN Foundation (Unknown); IESE Business School (Unknown); Uppsala University (Other); The Champalimaud Centre, Lisbon, Portugal (Unknown); Stockholm University (Other); University of Groningen, The Netherlands (Unknown); National Institute of Mental Health, Czech Republic (Other); European Association for Palliative Care (EAPC) (Unknown); Madopa (Unknown); Bispebjerg Hospital (Other); European Association of Neurological Associations (EFNA) (Unknown); 29k International AB (Unknown); Lung Alliance Netherlands (Unknown); European Psychiatric Association (Unknown); Norrsken Mind (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 18870; 2023-510488-36-01 (EU CTIS Number)
Record Dates: First submitted 2025-01-02; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); ALS (Amyotrophic Lateral Sclerosis); MS (Multiple Sclerosis); Major Depressive Disorder (MDD); Atypical Parkinson Disease
Keywords: psilocybin; therapy; palliative; care; palliative care; end-of-life distress; depression; psychological distress; psypal; copd; als; ms; apd; chronic obstructive pulmonary disorder; amyotrophic lateral sclerosis; multiple sclerosis; major depressive disorder; atypical parkinson disease; existential distress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Amyotrophic Lateral Sclerosis; Multiple Sclerosis; Depressive Disorder, Major; Parkinson Disease, Familial, Type 1; Depression

STUDY DESIGN:
Intervention Model Description: randomized double-blind low-dose controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate (15mg) and high dose (25mg) psilocybin group (Experimental): Patients assigned to this arm will first receive three prepration sessions followed by one moderate dose (15mg) of psilocybin. Patients will then receive two integration sessions and a high dose (25mg) of psilocybin. This is followed by three integration sessions.
  Interventions: Drug: Psilocybin therapy
- Low-dose (1mg) psilocybin group (Placebo Comparator): Patients assigned to this arm will first receive three prepration sessions followed by one low dose (1mg) of psilocybin. Patients will then receive two integration sessions and another low dose (1mg) of psilocybin. This is followed by three integration sessions.
  Interventions: Drug: Psilocybin therapy

INTERVENTIONS:
Drug: Psilocybin therapy — Psilocybin therapy consisting of three preparation, two dosing, and three integration sessions. All sessions will take place in a controlled, safety environment and supported by two study therapists

SUMMARY:
The goal of this clinical trial is to evaluate whether psilocybin therapy can effectively treat depression and psychological distress in adult patients with COPD, ALS, MS, or APD who have at least 6 months life expectancy. The main questions it aims to answer are:

* Can psilocybin therapy safely reduce depressive symptoms compared to low-dose control?
* Will the therapeutic effects be rapid and sustained over a 6-month period?

Researchers will compare patients receiving two escalating doses of psilocybin (15mg followed by 25mg) against those receiving two low doses (1mg) to see if the higher doses lead to greater improvements in depression, anxiety, demoralization, and quality of life.

Participants will:

* Attend three preparation sessions with psychotherapists (1-2 hours each)
* Undergo two supervised psilocybin dosing sessions (6-8 hours each)
* Complete five integration therapy sessions following the dosing sessions
* Participate in follow-up assessments at 6 weeks, 3 months, and 6 months
* Have access to a digital care platform and peer support groups during the 6-month follow-up period
* Optional: Control group participants may receive one high-dose psilocybin session (25mg) after the initial study period

DETAILED DESCRIPTION:
Rationale Patients with chronic obstructive pulmonary disorder (COPD), amyotrophic lateral sclerosis (ALS), multiple sclerosis (MS), or atypical and advanced Parkinsonian disorder (APD) often suffer from severe psychological distress with demoralization and death anxiety, which may culminate in to depressive disorder. Treatments of depression in palliative care currently involves psychotherapy and/or the use of antidepressants. However, these treatments have shown limited efficacy which urgently calls for new and innovative approaches. In recent years, a number of studies have shown very promising results of psilocybin therapy in alleviating psychological distress in patients with advanced cancer. The current study (PsyPal) aims to evaluate whether psilocybin therapy can also lead to rapid and sustained decreases in depressive symptoms, demoralization and other facets of psychological distress in patients who suffer from COPD, ALS, MS and APD.

Objective The primary objective of the PsyPal study is to assess the safety and efficacy of psilocybin therapy compared to low-dose control in reducing depressive symptoms in patients with COPD, ALS, MS, or APD. Secondary objectives of PsyPal are to assess change in clinical functioning, end-of-life anxiety, psychological/existential distress, health-related quality of life, and how it impacts caregiver 's health- and economic burden. The safety objective of PsyPal is to evaluate the difference in adverse events between high and low dose groups before, during and after the dosing session. Exploratory objectives include the investigation of psychological mechanism, subjective effects, biomarkers (EEG and blood-based), cost-effectiveness, and the usefulness of a digital care platform, with a mixed methods approach.

Main trial endpoints The main trial endpoint for PsyPal is the change in depression severity from baseline to 6 weeks after the second dose of psilocybin (high dose session). Adverse events and change in depression symptoms will also be assessed at 3- and 6-month follow-up to determine the safety and sustained effects of psilocybin therapy.

Secondary trial endpoints Secondary trial endpoints will be assessed at baseline and 6 weeks after the second dose of psilocybin. These include response rate, anxiety, demoralization, health-related quality of life, experiential avoidance, coping with illness, death anxiety, the wish to hasten death, self-compassion, spirituality, attachment, pain, healthcare resource use, blood-based biomarkers, and functional brain changes. Some secondary endpoints will also be assessed at the 3- and 6-month follow-up, including anxiety, demoralization, health-related quality of life, experiential avoidance, and coping with illness. These endpoints aim to improve our understanding of the effects of psilocybin therapy, how psilocybin therapy works, and to see which patients show the best response. Finally, changes in (religious/spiritual) beliefs/understandings and the experience(s) with psilocybin therapy will be assessed through in-depth qualitative interviews with patients that are conducted 6 weeks after the second dose of psilocybin.

Trial design PsyPal trial consists of a double-blind randomized low-dose controlled clinical trial with long term follow-up. Patients who are enrolled in the trial will be actively participating for ten weeks. After the primary endpoint, patients who received a low dose of psilocybin (1 mg) will be offered an optional single open label high-dose of psilocybin (25mg) together with three integration sessions. During long-term follow-up, patients will have access to a digital care platform and peer support groups.

Trial population The trial population in PsyPal consists of patients with COPD, ALS, MS, or APD and co-morbid depression. The main further inclusion criteria for participation are an age of 18 or higher, having an identified caregiver or support person, and a life expectancy of at least 6 months. The main exclusion criteria are current use of antipsychotic drugs, suicidal ideations, schizophrenia or other psychotic disorders, bipolar I/II disorder, other major neurological conditions, cardiovascular conditions, diabetes, and/or moderate to severe hepatic impairment (i.e., liver failure). Other exclusion criteria are a first-degree relative on the schizophrenia spectrum, other psychotic disorders, or bipolar I disorder.

Interventions

Patients will receive psilocybin therapy consisting of three phases; 1) preparation, 2) dosing, and 3) integration:

Preparation - The preparation phase consists of three psychotherapy sessions of 1-2 hours each. The purpose of these sessions is threefold: to build a therapeutic alliance between the patient and the therapist, to make a psychotherapeutic treatment plan for the patient using a process-based approach, and to educate patients about psilocybin's acute effects and how patients and therapists together can handle difficult experiences during the dosing sessions.

Dosing - The dosing phase of PsyPal starts 1-3 days after the last preparation session. It consists of two escalating dosing sessions of 6-8 hours each. The patient first receives a moderate dose of psilocybin (15mg). Two weeks later, the patient receives a high dose of psilocybin (25mg). Patients in the control group will receive two doses of psilocybin (1mg). All dosing sessions take place under supervision of two trained therapists within a treatment room specifically designed for psilocybin therapy and with a medical doctor on call.

Integration - The integration phase consists of five psychotherapeutic sessions of 1-2 hours each. There are two integration sessions following the first dosing session and three integration sessions following the second dosing session. The integration sessions are intended for further psychotherapeutic work, including working with the experience(s) that may have emerged during dosing sessions, and clinical assessment of the patient. Central topics may include the relationship with their life-limiting illness, death, meaning, sense of purpose, personal (religious/spiritual) beliefs, (social) relationships, and conflict resolution. The patient can also share thoughts and feelings about the PsyPal trial.

Long-term follow-up After the intervention, patients will be returned to regular care and followed for a period of 6 months, tracking usage of healthcare resources, the digital care platform, and peer support groups. Qualitative aspects of the intervention will be evaluated for patients, caregivers and therapists. Long-term safety data of psilocybin therapy will be collected for the four patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has to be diagnosed with one of the following four conditions, defined as:

   COPD i) Diagnosis by medical specialist ii) Postbronchodilator FEV1/FVC < 0,7 and FEV1 <80% pred iii) ≥ 40 years old iv) ≥ 10 years smoking

   ALS i) ALS according to Goldcoast criteria (Shefner et al, Clin Neurophysiol, 2020) ii) ALS-FRS-R subscores of minimum 1 in item 2, 3 and 8, subscore of minimum 2 in item 1, 4 and 10 and a subscore of minimum 3 in item 11 and 12

   MS i) Fulfilled diagnostic revised McDonald criteria for MS from 2017 (Thompson et al., 2018) ii) EDSS ≥ 1,0

   APD i) Advanced to Late-Stage Parkinson's Disease - patients with a diagnosis of Parkinson's Disease per the MDS clinical diagnosis criteria with evidence of motor and non-motor fluctuations ii) Diseases in the spectrum of Progressive supranuclear palsy (PSP), fulfilling possible and probable criteria, according to the MDS diagnostic criteria iii) Clinically Established and Clinically Probable Multiple System Atrophy (MSA) according to the MDS diagnostic criteria
2. Patient meets ICD-10 criteria for major depressive disorder documented through the com-pletion of the mood section of the Mini International Neuropsychiatric Interview by a screen-ing psychologist or physician.
3. Patient has a MADRS score of > 19.
4. Patient should have a life expectancy of at least 6 months (assessed by study physician).
5. Patient is at least 18 years of age.
6. Patient has an identified caregiver/support person. See specific conditions for Czechia in Appendix 5.
7. Patient is able to read and understand the informed consent and all scales used in a local language. For those with ALS, MS, or APD, competency is ensured via neurologist assessment, cognitive screening, caregiver support during screening and interactive approaches where the screening clinician ask the patient to explain their understanding of consent elements, re-explaining potentially misunderstood information.
8. Patient is able to and willing to adhere to study requirements, including attending all study visits, preparatory and follow-up sessions, and completing all study evaluations.
9. Patient is able to ingest capsules.

Exclusion Criteria:

1. Patient has used a psychedelic substance in the past 6 months (e.g., psilocybin, LSD, 5-MeO-DMT, DMT, ayahuasca or mescaline).
2. Patient is in active treatments for other psychiatric disorders, judged by the screening clinician to be a more significant clinical problem than depression / distress.
3. Patient meets ICD-10 criteria for schizophrenia spectrum or other psychotic disorders, including major depressive disorder with psychotic features (except substance/medication-induced or due to another medical condition) or bipolar I/II disorder.
4. Patients with any lifetime diagnosis of schizophrenia spectrum or other psychotic disorders.
5. Patient has a first-degree relative with schizophrenia spectrum, bipolar I disorder or other psychotic disorders (expect substance/medication-induced or due to another medical condition).
6. Patients with a pre-existing psychiatric condition judged to be incompatible with safe exposure to psilocybin therapy.
7. Significant suicide risk as defined by (1) suicidal ideation with intent to act (defined as ≥ 5 on MADRS item 10), (2) suicidal attempts within the past year, or (3) clinical assessment of significant suicidal risk during patient interview.
8. Patient meets ICD-10 criteria for active/current alcohol or drug use disorder.
9. Patient has ongoing treatment with antipsychotic drugs. Any prohibited agents must have been stopped at least 5x the elimination half-life of the specific drug at the time of baseline (see Appendix 1a for Prohibited medications).
10. Patient is unwilling or unable to pause formal psychotherapy (days 0-42).
11. Patient has neurological conditions (e.g., intracranial tumour, epilepsy, brain injuries, or other neurological disorders) expected by the PIs to conflict with the treatment / study protocol.
12. Disease-specific exclusion criteria:

    COPD: Unresolved exacerbation or pulmonary infection within last 4 weeks. ALS: Significant cognitive deficits (MoCa, see below). MS: Significant cognitive deficits (MoCa, see below), epilepsy or radiologically isolated syndrome.

    APD: Dementia (MoCa, see below), or Schwab and England ADL scale with scores > 80% in the best functional state.
13. Cardiovascular conditions: recent stroke (< 1 year from signing of ICF), recent myocardial infarction (< 1 year from signing of ICF), uncontrolled hypertension (blood pressure > 140/90 mmHg), clinically significant arrhythmia within 1 year of signing the ICF, or QTc prolongation exceeding 450ms (males) / 470ms (females).
14. Patient has moderate to severe hepatic impairment (Child-Pugh score ≥ 7).
15. Patient has insulin-dependent diabetes or who are taking oral hypoglycaemic agents and have a current risk of hypoglycaemia that would require medical intervention.
16. Patient has any physical or psychological symptoms, medications, blood test results or clinically significant findings at Screening or Baseline (based on the clinical judgement of clinical/medical study personnel) that would make a patient unsuitable for the study.
17. Patient has an allergy or intolerance to any of the materials contained in either drug product.
18. Cognitive and Neuropsychological assessment: Patients will be excluded if they score below mean minus 1.5 Standard Deviation according to normative age and scholarity adjusted data on the Montreal Cognitive Assessment (MoCA) assessment.
19. Recent (2 weeks) change or planned change in antidepressant medication during the intervention.
20. Women who are pregnant, intend to become pregnant during the study or who are currently nursing, or are unwilling to use Highly Effective Contraceptive Methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (MADRS) | Baseline (Day -14) to Primary Endpoint (Day 56)
  To examine medium/high-dose psilocybin therapy safety and efficacy in reducing symptoms of depression in patients with COPD, ALS, MS, or APD, compared to the low-dose control group.

SECONDARY OUTCOMES:
Response rate | Baseline (Day -14) to Primary Endpoint (Day 56)
  To determine the response rate to psilocybin therapy (≥50% reduction in MADRS)
End-of-life anxiety | Baseline (Day -14) to Primary Endpoint (Day 56)
  To evaluate the effect of psilocybin therapy on end-of-life anxiety
  - Death and Dying Distress Scale (DADDS)
Anxiety and depression (symptoms) | Baseline (Day -14) to Primary Endpoint (Day 56)
  To evaluate the effect of psilocybin therapy on symptoms of anxiety and depression
  - Hospital Anxiety and Depression Scale (HADS)
Demoralization | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on demoralization
  - Demoralization Scale-II (DS-II)
Impact on Quality of life | Baseline (Day -14) to Primary Endpoint (Day 56)
  To evaluate the effect of psilocybin therapy on quality of life
  - EQ-5D-5L
Caregiver burden | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on caregiver burden
  - Zarit Burden Interview (ZBI-7)
Daily functioning in COPD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on daily function in patients with COPD.
  - CODP Assessment Test (CAT)
Health-related quality of life in COPD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on health-related quality of life in patients with COPD.
  - St. George's Respiratory Questionnaire (SGRQ-C)
Health-related quality of life in ALS | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on quality of life in patients with ALS.
  - Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALS-AQ-5)
Functional status in ALS | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on functional status in patients with ALS
  - ALS Functional Rating Scale Revised (ALS-FRS-R)
Health-related quality of life in MS | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on health-related quality of life in patients with MS.
  - Expanded Disability Status Scale (EDSS)
Health-related quality of life in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on health-related quality of life in patients with APD.
  - Parkinson's Disease Questionnaire (PDQ-8)
Motor and non-motor symptoms in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on (non-)motor symptoms in patients with APD.
  - Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS, parts I, II, and III)
Functional magnetic resonance imaging (fMRI) in APD | Baseline (Day -14) to one week after Dose 2 (Day 21)
  At the Champalimaud Foundation in Lisbon, structural and functional magnetic resonance imaging (MRI) will be conducted in patients with APD. Changes in brain volume and tissue microstructures (with fractional anisotropy and diffusivity) will be computed. Changes in whole brain resting-state functional connectivity will be additionally computed using the BOLD response. The structural and function MRI protocol consists of 3D T1-weighted, T2/PD-weighted, FLAIR, T2*, diffusion tensor, and blood-oxygen-level-dependent (BOLD) imaging.
Incidence, severity, and frequency of (serious) adverse events following psilocybin therapy | Baseline (Day -14), Dose 1 (Day 0), Integration 1 (Day 1), Integration 2 (Day 7), Dose 2 (Day 14), Integration 3 (Day 15), Integration 4 (Day 21), Integration 5 (Day 28), Primary endpoint (Day 56), Open label dose (Day 62), 3- and 6-month follow-up
  The reporting of (serious) adverse events by using MedDRA version 27.0 during the clinical trial.

OTHER OUTCOMES:
Experiential avoidance | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on experiential avoidance
  - Brief Experiential Avoidance Questionnaire (BEAQ)
Coping | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on coping with a chronic illness
  - BRIEF-COPE questionnaire
The wish to hasten death | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on the wish to hasten death
  - Scheduled Attitudes towards Hastened Death (SAHD)
Self-compassion | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on self-compassion
  - Self-Compassion Scale Short-Form (SCS-SF)
Attachment | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on attachment
  - Experientience in Close Relationships (ECR)
Pain perception | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on pain perception
  - Numeric Rating Scale
Spiritual well-being | Baseline to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on spiritual well-being
  - Functional Assessment of Chronic Illness Therapy - Spiritual well-being 12 (FACIT-Sp-12)
Mystical experience | Dosing session 1 (Day 0) and Dosing session 2 (Day 14)
  To assess whether psilocybin induces a mystical experience using the Mystical Experience Questionnaire (MEQ-30) and explore how it relates to antidepressant efficacy and other related outcome measures (e.g., anxiety, death anxiety, demoralization).
Emotional breakthrough | Dosing session 1 (Day 0) and Dosing session 2 (Day 14)
  To assess whether psilocybin results in an emotional breakthrough using the Emotional Breakthrough Inventory (EBI) and explore how it relates to antidepressant efficacy and other related outcome measures (e.g., anxiety, death anxiety, demoralization).
Challenging experiences | Dosing session 1 (Day 0) and Dosing session 2 (Day 14)
  To assess whether psilocybin induces challenging experiences using the Challenging Experience Questionnaire (CEQ) and explore how it relates to antidepressant efficacy and other related outcome measures (e.g., anxiety, death anxiety, demoralization).
Experience of music during dosing sessions | Dose 1 (Day 0) and Dose 2 (Day 14)
  To assess how study participants experience during the dosing session and explore how it relates to antidepressant efficacy and other related outcome measures (e.g., anxiety, death anxiety, demoralization).
Brain function | Baseline (Day -14), one day after Dose 1 (Day 1), and one day after Dose 2 (Day 15)
  To assess whether there are changes in prefrontal theta activity following psilocybin therapy brain using electroencephalogrphy (EEG) in patients with COPD and MS. Time-frequency analyses will be conducted and various ERP components will be examined, particularly the LPP, N2b, and P300. Other exploratory measures include frontal alpha asymmetry, frontoparietal alpha and theta power, ECG-derived average heart rate and heart rate variability occipital alpha asymmetry, parieto-occipital alpha power, Lempel-Ziv Complexity, and State-Space Entropy .
  The EEG assessments include a resting-state scan (10 minutes) and an emotional reactivity scan (10 minutes), where patients are presented with neutral (n=24), negative (n=24), and positive (n=24) stimuli. Each stimulus is presented for 2 seconds followed by a question about the emotional intensity.
Blood-based biomarkers | Baseline (Day -14) to Dose 2 (Day 14) and primary endpoint (Day 56)
  To assess whether there are changes in blood-based biomarkers following psilocybin therapy by using serum and plasma analysis of several different neuroendocrine (cortisol, prolactin, oxytocin, ACTH), inflammatory (CRP, IL-1 beta, IL-6, and TNF-alpha), neurotrophic (brain-derived neurotrophic factor and Val66Met), and neurological (neurofilaments) biomarkers. Gene expression in intracellular RNA in whole blood will also be analyzed as well as psilocin concentration in plasma during dosing sessions.
Cost-effectiveness | Baseline (Day -14) to Primary Endpoint (Day 56)
  To evaluate the cost-effectiveness of psilocybin therapy, taking into account health gains for patients and caregivers as well as costs of the therapy and use of societal resources.
Long-term positive and negative effects | Baseline (Day -14) to Primary Endpoint (Day 56) and 3-month (Day 104) and 6-month follow-up (Day 194)
  To monitor long-term positive and negative effects of psilocybin therapy through the evaluation of quantitative and qualitative methods
Verbal learning and memory in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on verbal learning and memory in patients with APD.
  - Rey Auditory Verbal Learning Test
Working memory and attention in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on working memory and attention in patients with APD.
  - Letters and Numbers Sequence
Cognitive flexibility in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on cognitive flexibility in patients with APD.
  - Trail Making Test
Executive function, lexical retrieval, and processing speed in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on executive function, lexical retrieval, and processing speed in patients with APD.
  - Verbal Fluency
Sustained attention and working memory in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on attention and working memory in patients with APD.
  - Digit Span
Processing speed, working memory, sustained attention, visual-motor coordination, and executive function in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on processing speed, working memory, sustained attention, visual-motor coordination, and executive function in patients with APD.
  - Digit Symbol Substitution Test
Reading skills in APD | Baseline (Day -14) to Primary Endpoint (Day 56)
  To assess the impact of psilocybin therapy on reading skills in patients with APD.
  - Irregular Word Reading Test
Optional: qualitative interviews (patients) | After Primary Endpoint (Day 56)
  Online or in-person semi-structured interviews to explore lived experiences of psilocybin therapy in patients with COPD, ALS, MS, or APD.
Optional: focus group (patients) | At the end of Long-Term Follow-Up (Day 194)
  Online focus groups to exchange experiences of psilocybin therapy with peers
Optional: journaling (patients) | Continuous during clinical trial
  Patient are asked to reflect on their experience with psilocybin therapy through a journal during the clinical trial.
Optional: focus groups (therapists) | At the end of Long-Term Follow-Up (Day 194)
  Online focus groups with therapists to explore their perspective on psilocybin therapy
Optional: journaling (therapists) | Baseline to 3-month and 6-month follow-up
  Therapists are asked to reflect on their experience with psilocybin therapy through a journal during the clinical trial.
Optional: focus group (caregivers) | After Primary Endpoint (Day 56) and at the end of Long-Term Follow-Up (Day 194)
  Online focus groups with caregivers to explore their perspective on psilocybin therapy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official website for PsyPal — https://palliativeprojects.eu/psypal/